CLINICAL TRIAL: NCT01275066
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multinational Clinical Study to Evaluate the Efficacy and Safety of 2.0 mg/kg/Week and 2.0 mg/kg/Every Other Week BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Brief Title: A Double-Blind Study to Evaluate the Efficacy and Safety of BMN 110 in Patients With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR-004; 2010-020198-18 (EudraCT Number); 10/H1306/87 (Other: National Research Ethics Service); 18972/0213/001-0001 (Other: Medicines and Healthcare Products Regulatory Agency); 2011_038#B201129 (Other: Medical Ethics Review Committee (METC)); 145240 (Other: Health Canada); 2011-01-09 (Other: Committee for the Protection of Personnes); 20110012889 (Other: Korean Food & Drug Administration (KFDA)); 0999935174 (Other: Taiwan FDA)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2014-07-07 (Estimated); Status verified 2014-06

CONDITIONS: MPS IV A
Keywords: Mucopolysaccharidosis IV type A; MPS IV Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — Chondroitinsulfatases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BMN 110 Weekly (Experimental)
  Interventions: Drug: BMN 110 Weekly
- BMN 110 Every Other Week (Experimental)
  Interventions: Drug: BMN 110 Every Other Week

INTERVENTIONS:
Drug: BMN 110 Weekly — BMN 110 Weekly: Intravenous infusion of BMN 110 at a dose of 2.0 mg/kg administered over a period of approximately 4 hours once a week.
  Other Names: recombinant human N-acetylgalactosamine-6-sulfatase; rhGALNS
  Arms: BMN 110 Weekly
Drug: Placebo — Intravenous infusion of placebo solution at a volume equivalent to that needed for 2.0 mg/kg dose of BMN 110 administered over a period of approximately 4 hours once a week.
  Arms: Placebo
Drug: BMN 110 Every Other Week — BMN 110 Every Other Week: Intravenous infusion of BMN 110 at a dose of 2.0 mg/kg administered over a period of approximately 4 hours every other week and infusions of placebo on alternating weeks.
  Other Names: recombinant human N-acetylgalactosamine-6-sulfatase; rhGALNS
  Arms: BMN 110 Every Other Week

SUMMARY:
This Phase 3 study will evaluate the efficacy and safety of 2.0 mg/kg/week BMN 110 and 2.0 mg/kg/every other week BMN 110 in patients with mucopolysaccharidosis IVA (Morquio A Syndrome).

There is currently no standard accepted treatment for MPS IVA other than supportive care. Enzyme replacement therapy (ERT) may be a potential new treatment option for MPS IVA patients. BMN 110 is administered to MPS IVA patients by IV infusion, allowing cellular uptake by the mannose-6-phosphate receptor and transportation to the lysosomes.

This enzyme uptake into the lysosomes is hypothesized to promote increased catabolism of keratan sulfate (KS) in tissue macrophages, hyaline cartilage, other connective tissues, and heart valve, and reduce the progressive accumulation of KS which is responsible for the clinical manifestations of the disorders.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 years of age.
* Documented clinical diagnosis of MPS IVA based on clinical signs and symptoms of MPS IVA and documented reduced fibroblast or leukocyte GALNS enzyme activity or genetic testing confirming diagnosis of MPS IVA.
* Willing and able to provide written, signed informed consent, or in the case of patients under the age of 18 (or 16 years, depending on the region), provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Must meet the study entrance requirements for the 6-minute walk test.
* Sexually active patients must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study.

Exclusion Criteria:

* Previous hematopoietic stem cell transplant (HSCT).
* Previous treatment with BMN 110.
* Has known hypersensitivity to any of the components of BMN 110.
* Major surgery within 3 months prior to study entry or planned major surgery during the 24-week treatment period.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Concurrent disease or condition, including but not limited to symptomatic cervical spine instability, clinically significant spinal cord compression, or severe cardiac disease that would interfere with study participation or safety as determined by the Investigator.
* Any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lounsbury, Study Director — BioMarin Pharmaceutical
Locations (28):
- United States (6):
  - Oakland, California
  - Wilmington, Delaware
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - New York, New York
  - Seattle, Washington
- Córdoba, Argentina
- Brazil (2):
  - Campina Grande
  - Porto Alegre
- Canada (3):
  - Montreal
  - Sherbrooke
  - Toronto
- Bogotá, Colombia
- Copenhagen, Denmark
- France (2):
  - Lyon
  - Paris
- Mainz, Germany
- Monza, Italy
- Tokyo, Japan
- Amsterdam, Netherlands
- Coimbra, Portugal
- Doha, Qatar
- Riyadh, Saudi Arabia
- Seoul, South Korea
- Taipei, Taiwan
- United Kingdom (3):
  - Birmingham
  - London
  - Manchester

REFERENCES:
- [Derived] Schweighardt B, Tompkins T, Lau K, Jesaitis L, Qi Y, Musson DG, Farmer P, Haller C, Shaywitz AJ, Yang K, O'Neill CA. Immunogenicity of Elosulfase Alfa, an Enzyme Replacement Therapy in Patients With Morquio A Syndrome: Results From MOR-004, a Phase III Trial. Clin Ther. 2015 May 1;37(5):1012-1021.e6. doi: 10.1016/j.clinthera.2014.11.005. Epub 2014 Dec 6. PMID 25487082
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN110 2.0 mg/kg/Qow: Intravenous infusion of BMN 110 at a dose of 2.0 mg/kg administered over a period of approximately 4 hours every other week and infusions of placebo on alternating weeks.
- BMN110 2.0 mg/kg/Week: Intravenous infusion of BMN 110 at a dose of 2.0 mg/kg administered over a period of approximately 4 hours once a week.
Period: Overall Study
Arm/Group | Placebo | BMN110 2.0 mg/kg/Qow | BMN110 2.0 mg/kg/Week
Started | 60 | 59 | 58
Treated | 59 | 59 | 58
Completed | 59 | 59 | 57
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Not Diagnosed w/ Disease | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BMN110 2.0 mg/kg/Qow | BMN110 2.0 mg/kg/Week | Total
Number analyzed (Participants) | 59 | 59 | 58 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (11.30) | 15.3 (10.79) | 13.1 (8.10) | 14.5 (10.16)
Age, Customized [Number; unit: participants]
  5 - 11 years | 30 | 31 | 32 | 93
  12 - 18 years | 15 | 16 | 16 | 47
  >= 19 years | 14 | 12 | 10 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 25 | 32 | 89
  Male | 27 | 34 | 26 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 9 | 38
  Not Hispanic or Latino | 46 | 43 | 49 | 138
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 15 | 14 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 44 | 35 | 36 | 115
  Other | 4 | 7 | 6 | 17
Region of Enrollment [Number; unit: participants]
  Argentina | 1 | 1 | 0 | 2
  Brazil | 6 | 10 | 5 | 21
  Canada | 4 | 5 | 5 | 14
  Colombia | 2 | 2 | 2 | 6
  Denmark | 0 | 0 | 1 | 1
  France | 7 | 5 | 8 | 20
  Germany | 4 | 5 | 1 | 10
  Italy | 4 | 4 | 2 | 10
  Japan | 0 | 4 | 2 | 6
  Korea, South | 3 | 1 | 3 | 7
  Netherlands | 1 | 2 | 3 | 6
  Portugal | 2 | 1 | 0 | 3
  Qatar | 1 | 0 | 1 | 2
  Saudi Arabia | 2 | 1 | 4 | 7
  Taiwan | 1 | 3 | 1 | 5
  United Kingdom | 9 | 4 | 10 | 23
  United States | 12 | 11 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Endurance as Measured by the 6-minute Walk Test
Time Frame: Baseline to Week 24
Population: Intention to treat (all patients receiving at least one dose of study drug). Two missing outcomes at Week 24 were imputed using method of multiple imputation.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | BMN110 2.0 mg/kg/Qow | BMN110 2.0 mg/kg/Week
Number analyzed (Participants) | 59 | 59 | 58
meters
  Baseline | 211.9 (69.88) | 205.7 (81.19) | 203.9 (76.32)
  Week 24 | 225.4 (83.22) | 219.9 (87.60) | 240.0 (86.61)
  Change from Baseline to Week 24 | 13.5 (50.63) | 14.2 (40.82) | 36.0 (58.11)
Statistical Analysis 1: Comparison: Placebo vs BMN110 2.0 mg/kg/Week; Test type: Superiority or Other; p = 0.0174, ANCOVA — Hochberg multiplicity adjustment - results considered statistically significant if both of p-values are p<0.05 or either of p-values is p<0.025; ANCOVA of change from baseline with treatment, age group, baseline 6MWT category as covariates; Mean Difference (Final Values) = 22.5, Standard Error of Mean 9.35
Statistical Analysis 2: Comparison: Placebo vs BMN110 2.0 mg/kg/Qow; Test type: Superiority or Other; p = 0.9542, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA of change from baseline with treatment, age group, baseline 6MWT category as covariates; Mean Difference (Final Values) = 0.5, Standard Error of Mean 9.29

2. Secondary Outcome: Change From Baseline in Endurance as Measured by the 3-minute Stair Climb Test
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: stairs/minute
Arm/Group | Placebo | BMN110 2.0 mg/kg/Qow | BMN110 2.0 mg/kg/Week
Number analyzed (Participants) | 59 | 59 | 58
stairs/minute
  Baseline | 30.0 (14.05) | 27.1 (15.80) | 29.6 (16.44)
  Week 24 | 33.6 (18.36) | 30.4 (17.77) | 34.3 (18.70)
  Change from Baseline to Week 24 | 3.6 (8.51) | 3.2 (10.29) | 4.7 (7.99)
Statistical Analysis 1: Comparison: Placebo vs BMN110 2.0 mg/kg/Week; Test type: Superiority or Other; p = 0.4935, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA of change from baseline with treatment, age group, baseline 6MWT category, and baseline 3MSCT as covariates; Mean Difference (Final Values) = 1.1, Standard Error of Mean 1.66
Statistical Analysis 2: Comparison: Placebo vs BMN110 2.0 mg/kg/Qow; Test type: Superiority or Other; p = 0.7783, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA of change from baseline with treatment, age group, baseline 6MWT category, and baseline 3MSCT as covariates; Mean Difference (Final Values) = -0.5, Standard Error of Mean 1.66

3. Secondary Outcome: Percent Change From Baseline in Urine Keratan Sulfate Normalized for Urine Creatinine
Time Frame: Baseline to Week 24
Population: Intention to treat (all patients receiving at least one dose of study drug). Nine missing outcomes at Week 24 were imputed using method of multiple imputation.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | BMN110 2.0 mg/kg/Qow | BMN110 2.0 mg/kg/Week
Number analyzed (Participants) | 59 | 59 | 58
percent change | -3.6 (27.41) | -35.3 (20.74) | -43.7 (22.29)
Statistical Analysis 1: Comparison: Placebo vs BMN110 2.0 mg/kg/Week; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA of change from baseline with treatment, age group, baseline 6MWT category, and baseline uKS normalized for creatinine, as covariates; Mean Difference (Final Values) = -40.7, Standard Error of Mean 4.20
Statistical Analysis 2: Comparison: Placebo vs BMN110 2.0 mg/kg/Qow; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -30.2, Standard Error of Mean 4.19

ADVERSE EVENTS:
Time Frame: Study Period, through 24 weeks
Description: Treatment Emergent Events Only
Arm/Group | Placebo | BMN110 2.0 mg/kg/Qow | BMN110 2.0 mg/kg/Week
Serious Adverse Events (participants affected / at risk) | 2/59 | 4/59 | 9/58
Other Adverse Events (participants affected / at risk) | 57/59 | 59/59 | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | BMN110 2.0 mg/kg/Qow (N=59) | BMN110 2.0 mg/kg/Week (N=58)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Suture removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | BMN110 2.0 mg/kg/Qow (N=59) | BMN110 2.0 mg/kg/Week (N=58)
Mitral valve incompetence (Cardiac disorders) | 4 (4) | 3 (3) | 3 (3)
Pulmonary valve incompetence (Cardiac disorders) | 2 (2) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 6 (7) | 2 (6) | 3 (8)
Tricuspid valve incompetence (Cardiac disorders) | 3 (3) | 7 (7) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 5 (6) | 8 (11) | 3 (3)
Corneal opacity (Eye disorders) | 1 (1) | 0 (0) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 8 (14) | 14 (23)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 4 (4) | 9 (22)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 12 (14) | 12 (14)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (13) | 14 (22) | 18 (37)
Vomiting (Gastrointestinal disorders) | 21 (42) | 21 (44) | 25 (60)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 3 (3)
Chills (General disorders) | 1 (1) | 6 (7) | 6 (7)
Device occlusion (General disorders) | 1 (1) | 2 (2) | 3 (4)
Fatigue (General disorders) | 15 (24) | 8 (10) | 9 (17)
Infusion site extravasation (General disorders) | 2 (2) | 4 (4) | 2 (2)
Infusion site pain (General disorders) | 0 (0) | 4 (7) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 4 (6) | 1 (1)
Puncture site pain (General disorders) | 2 (2) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 17 (29) | 22 (35) | 25 (47)
Hypersensitivity (Immune system disorders) | 1 (1) | 4 (7) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 5 (5)
Gastroenteritis (Infections and infestations) | 4 (4) | 8 (10) | 7 (8)
Influenza (Infections and infestations) | 3 (4) | 5 (5) | 2 (3)
Nasopharyngitis (Infections and infestations) | 9 (12) | 12 (13) | 10 (11)
Otitis media (Infections and infestations) | 4 (4) | 5 (5) | 8 (9)
Pharyngitis (Infections and infestations) | 7 (7) | 3 (3) | 4 (4)
Rhinitis (Infections and infestations) | 6 (8) | 4 (8) | 5 (8)
Upper respiratory tract infection (Infections and infestations) | 9 (14) | 10 (13) | 10 (15)
Viral infection (Infections and infestations) | 1 (1) | 6 (6) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 3 (5) | 4 (5) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 2 (5) | 3 (4) | 2 (2)
Blood pressure systolic increased (Investigations) | 2 (5) | 3 (16) | 1 (1)
Body temperature increased (Investigations) | 2 (10) | 2 (2) | 4 (24)
Oxygen saturation decreased (Investigations) | 6 (19) | 7 (8) | 6 (10)
Respiratory rate increased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (27) | 9 (14) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (17) | 7 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 3 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 5 (6)
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (13) | 14 (24) | 9 (16)
Dizziness (Nervous system disorders) | 3 (3) | 4 (6) | 7 (10)
Headache (Nervous system disorders) | 21 (38) | 24 (52) | 24 (69)
Hyperreflexia (Nervous system disorders) | 3 (6) | 1 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (6)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (28) | 17 (29) | 16 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (8) | 7 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 5 (7) | 5 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (12) | 12 (14)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (9) | 5 (5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (7) | 6 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 3 (5)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 5 (7)
Hot flush (Vascular disorders) | 1 (1) | 4 (6) | 3 (3)
Hypertension (Vascular disorders) | 4 (13) | 4 (18) | 3 (6)
Hypotension (Vascular disorders) | 1 (1) | 2 (3) | 3 (3)
Poor venous access (Vascular disorders) | 4 (8) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less